CLINICAL TRIAL: NCT03943680
Title: Clinical Behavior and Molecular Pathways of PRGF in Post-extraction Sockets
Brief Title: Plasma Rich in Growth Factors in Post-extraction Sockets
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Collaborators: BTI Biotechnology Institute (Unknown)
Responsible Party: Principal Investigator, Pablo Galindo-Moreno, Professor, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1962-N-18
Record Dates: First submitted 2019-05-07; First posted 2019-05-09 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Tooth Extraction; Dental Implants
Keywords: Tooth extraction; Socket regeneration; Dental Implants

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PRGF (Experimental): Post-extraction socket grafted with PRGF-Endoret
  Interventions: Device: PRGF
- ABB (Active Comparator): Post-extraction socket grafted with anorganic bovine bone (ABB)
  Interventions: Device: ABB

INTERVENTIONS:
Device: PRGF — After tooth extraction, the socket will be grafted with PRGF-Endoret
  Other Names: PRGF-Endoret
  Arms: PRGF
Device: ABB — After tooth extraction, the socket will be grafted with Geistlich Bio-Oss® Collagen
  Other Names: Geistlich Bio-Oss® Collagen
  Arms: ABB

SUMMARY:
The purpose of this study is to compare the clinical success, radiographical volume maintenance and histological bone regeneration after using either a bovine bone xenograft or an autogenous platelet rich plasma enrich in growth factors, known as Endoret®-PRGF®.

ELIGIBILITY:
Inclusion Criteria:

* Upper or lower premolar or molar tooth in need of extraction and later restoration by dental implant.
* Adjacent and opposing natural teeth present and healthy.
* At least 3 mm from the tip of the dental root to the maxillary sinus or the inferior alveolar canal.

Exclusion Criteria:

* Active local infection.
* Uncontrolled diabetes mellitus.
* Long term (>10 years) use of oral bisphosphonates.
* Use of intravenous bisphosphonates.
* Recent use (<3 months) of antibiotics, antiinflammatories or analgesics drugs.
* Pregnancy.
* Smokers of more than 10 cigarettes per day.
* Any oral pathology that needs to be treated before tooth extraction, particularly the presence of more than 25% of sites with bleeding on probing.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2024-11-18 (Actual); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Alveolar bone change in Cone Beam Computerized Tomography | Baseline and 4 months
  Volumetric change in the alveolar bone from immediately after tooth extraction to immediately before implant placement (4 months after the extraction and grafting of the socket)

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Galindo-Moreno, DDS, PhD, Principal Investigator — Universidad de Granada
Locations (1):
- Facultad de Odontología, Granada, Granada, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Anitua E, Murias-Freijo A, Alkhraisat MH, Orive G. Clinical, radiographical, and histological outcomes of plasma rich in growth factors in extraction socket: a randomized controlled clinical trial. Clin Oral Investig. 2015 Apr;19(3):589-600. doi: 10.1007/s00784-014-1278-2. Epub 2014 Jul 8. PMID 24998770